CLINICAL TRIAL: NCT04179682
Title: The Pilot Study of Constraint Induced Movement Therapy(CIMT） Intervention in Children With Hemiplegic Cerebral Palsy After Botulism Toxin Injection in Preschool Education
Brief Title: A Pilot Study of Constraint Induced Movement Therapy in Preschool Cerebral Palsy After Botulism Toxin Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 130210
Record Dates: First submitted 2019-11-21; First posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Cerebral Palsy, Spastic; Rehabilitation
Keywords: cerebral palsy; constraint-induced movement therapy; botulinum toxin; rehabilitation; occupational therapy
MeSH Terms: conditions — Cerebral Palsy | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4-week 2-hours/day CIMT program (Active Comparator): a 4-week 2-hours/day constraint program, total 40 hours CIMT, in preschool education.
  Interventions: Procedure: 40-hour constraint-induced movement therapy
- 2-week 4-hours/day CIMT program (Active Comparator): one was a 2-week 4-hours/day constraint program, total 40 hours CIMT, in preschool education.
  Interventions: Procedure: 40-hour constraint-induced movement therapy

INTERVENTIONS:
Procedure: 40-hour constraint-induced movement therapy — Participants were randomly allocated to 1 of 2 CIMT programs (40 hours): a 2-week 4-hours/day CIMT program and a 4-week 2-hours/day CIMT program. One CIMT program was performed 1 month after a BoNT-A injection, and then the second program was implemented with the next injection.

SUMMARY:
To establish a pilot randomized, crossover study on applying 2 constraint-induced movement therapy (CIMT) interventions in children with hemiplegic cerebral palsy after botulinum toxin injection during preschool education.

DETAILED DESCRIPTION:
This study was designed to be a pilot study on the use of 4-week 2-hours/day and 2-week 4-hours/day CIMT interventions in children with hemiplegic CP after a BoNT-A injection in preschool education, and compared the effects and psychological stress of CP children relative to the 2 CIMT programs.

ELIGIBILITY:
Inclusion Criteria:

hemiplegic or quadriplegic CP children were under a regular rehabilitation program with BoNT-A injections. They were classified as Gross Motor Function Classification System level I and II, aged between 3 and 6 years old, with at least below average mentality, and were in mainstream preschool education; the extension of their hemiplegic wrist and metaphalangeal joint was greater than 10 degrees.

Exclusion Criteria:

Children were excluded if they (a) could not understand or cooperate with the CIMT program, (b) had joint contracture of an upper limb, and (c) could not actively extend their hemiplegic wrist.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2019-02-10 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
change of Modified Ashworth Scale(MAS) | 1 month after Botox injection, shortly after CIMT intervention, 2 months after CIMT, and 4 months after CIMT
  change of spasticity, from 0 to 4, higher scores mean a worse outcome.
change of Visual-motor integration in Peabody-Developmental Motor Scales(PDMSⅡ) | 1 month after Botox injection, shortly after CIMT intervention, 2 months after CIMT, and 4 months after CIMT
  hand function, from 0 to 144, higher scores mean a better outcome.
Change of grasping in Peabody-Developmental Motor Scales(PDMSⅡ) | 1 month after Botox injection, shortly after CIMT intervention, 2 months after CIMT, and 4 months after CIMT
  hand function. from 0 to 52, higher scores mean a better outcome.
Change of Chinese Version of Pediatric Evaluation of Disability Inventory( PEDI-C) | 1 month after Botox injection, shortly after CIMT intervention, 2 months after CIMT and 4 months after CIMT
  ADL, from 0 to 73, higher scores mean a better outcome.
Change of GAS(goal attainment scale) | 1 month after Botox injection, 2 months after CIMT and 4 months after CIMT
  GAS included 2 playing goals and 2 self-care goals.The goals were decided by the occupation therapist, the preschool teacher and the major caregiver. From (-2) to 2, higher scores mean a better outcome.
Change of Caregiver-Teacher Report Form (C-TRF)-Diagnostic scale of the Achenbach System of Empirically-Based Assessment (ASEBA) | 1 month after Botox injection, shortly after CIMT intervention, 2 months after CIMT and 4 months after CIMT
  From 0 to 14, higher scores mean a worse outcome.
Change of Statistical Manual (DSM)-oriented scale of the Achenbach System of Empirically-Based Assessment (ASEBA) | 1 month after Botox injection, shortly after CIMT intervention, 2 months after CIMT and 4 months after CIMT
  From 0 to 14, higher scores mean a worse outcome.

IPD SHARING:
Plan to Share IPD: No